CLINICAL TRIAL: NCT06055491
Title: Effect of Vitamin D3 Combined With Extensor Muscle Strengthening Exercise in Lateral Epicondylitis of Elbow: a Randomized Controlled Trial
Brief Title: Vitamin D3 Combined With Strengthening Exercise for Lateral Epicondylitis of Elbow
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Jung-Taek Hwang, Professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-07-018-001
Record Dates: First submitted 2023-09-15; First posted 2023-09-26 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Lateral Epicondylitis of Elbow
Keywords: Vitamin D3 injection; extensor strengthening exercise with counterforce brace; plasma Vitamin D3 level; visual analog scale of pain (VAS); Mayo Elbow Performance Score (MEPS); sonographic evaluation
MeSH Terms: conditions — Tennis Elbow | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Study group: Vitamin D3 injection at ilsilateral deltoid muscle and extensor muscle strengthening exercise with counterforce brace for lateral epicondylitis of elbow Control group: Saline injection at ilsilateral deltoid muscle and extensor muscle strengthening exercise with counterforce brace for lateral epicondylitis of elbow
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: An independent nurse uses a random sequence generator and allocates the participants into the two groups. Participant, investigator and outcomes assessor were blinded of participants' information
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D3 injection (Experimental): 1.0mL Vitamin D3 injection at ilsilateral deltoid muscle and extensor muscle strengthening exercise with counter force brace in lateral epicondylitis of elbow
  Interventions: Drug: Vitamin D3 or Saline injection at ipsilateral deltoid muscle
- Saline injection (Placebo Comparator): 1.0mL saline injection at ilsilateral deltoid muscle and extensor muscle strengthening exercise with counter force brace in lateral epicondylitis of elbow
  Interventions: Drug: Vitamin D3 or Saline injection at ipsilateral deltoid muscle

INTERVENTIONS:
Drug: Vitamin D3 or Saline injection at ipsilateral deltoid muscle — study group: 1.0mL Vitamin D3 injection control group: 1.0mL saline injection
  Other Names: extensor muscle strengthening exercise with counterforce brace

SUMMARY:
The goal of this study is to verify the effect of vitamin D3 combined with extensor muscle strengthening exercise in lateral epicondylitis of elbow Are there significant differences in the improvement of functional scores between the study and control groups? Are there significant differences in the improvement of sonographic findings and blood D3 levels between the study and control groups? Participant will underwent D3 injection or saline injection and extensor muscle strengthening exercise with counter force brace. All the participant will undergo functional scoring, sonographic examination and blood D3 level testings until 6 months after initial visit.

ELIGIBILITY:
Inclusion Criteria:

* lateral epicondylitis(LE) of elbow symptoms that persisted of increased for more than 3 months in which LE was defined as pain on the lateral side of the elbow and pain at the lateral epicondyle upon direct palpation and during resisted dorsiflexion of the wrist

Exclusion Criteria:

* younger than 20 years
* history of ipsilateral elbow surgery
* common extensor tendon tears more than 30% in depth
* inflammatory diseases (rheumatoid arthritis, psoriatic arthritis, etc)
* osteoarthritis with a limitation of range of motion (flexion contracture >30 degree and further flexion < 100 degree)
* neurological deficits in the ipsilateral upper limb,and follow-ups less than 24 weeks

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
visual analog scale of pain (VAS) | initial, Week 4, 12, 24
  0-10, 0: no pain, 10: very severe pain

SECONDARY OUTCOMES:
Patient's satisfaction | initial, Week 4, 12, 24
  0-10, 0: not satisfied, 10: very much satisfied
Mayo Elbow Performance Score (MEPS) | initial, Week 4, 12, 24
  0-100: higher score mean a better outcome
Grip power (attected/nonaffected) | initial, Week 4, 12, 24
  Newton/Newton
plasma Vitamin D level | initial, Week 4, 12, 24
  ng/mL
sonographic evaluation | initial, Week 4, 12, 24
  common extensor

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Taek Hwang, MD, PhD, Principal Investigator — Hallym University Medical Center
Locations (1):
- Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No
Our IRB does not permit

REFERENCES:
- [Result] Shim BJ, Seo EM, Hwang JT, Kim DY, Yang JS, Seo SJ, Hong MS. Comparison of the effectiveness of extensor muscle strengthening exercise by itself, exercise with polydeoxyribonucleotide injection, and exercise with extracorporeal shockwave therapy in lateral epicondylitis: a randomized controlled trial. Clin Shoulder Elb. 2021 Dec;24(4):231-238. doi: 10.5397/cise.2021.00290. Epub 2021 Nov 26. PMID 34823312